CLINICAL TRIAL: NCT02441439
Title: To Compare the Efficacy of I.V 200 mg Iron Sucrose and 500 mg Iron Sucrose to Treat Anemia in Pregnancy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The investigators decided not to proceed with this study
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, enav yefet, MD/PhD, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0036-15
Record Dates: First submitted 2015-05-06; First posted 2015-05-12 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Pregnancy
MeSH Terms: interventions — Ferric Oxide, Saccharated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iron sucrose 200 mg (Other): first arm will be treated with iron sucrose 200 mg 2-3 times a week
  Interventions: Dietary Supplement: Iron sucrose 200 mg
- Iron sucrose 500 mg (Active Comparator): Second arm will be treated with iron sucrose 500 mg once a week
  Interventions: Dietary Supplement: Iron sucrose 500 mg

INTERVENTIONS:
Dietary Supplement: Iron sucrose 200 mg — I.V Iron sucrose 200 mg 2-3 times per week. Each time for 20-30 minutes
  Arms: Iron sucrose 200 mg
Dietary Supplement: Iron sucrose 500 mg — I.V Iron sucrose 500 mg once per week. Each time for 3.5 hours
  Arms: Iron sucrose 500 mg

SUMMARY:
This study is aimed to compare the efficacy of 2 doses of iron sucrose given intravenously - 200 mg versus 500 mg.

DETAILED DESCRIPTION:
Anemia is common during pregnancy. It is associated with maternal and neonatal complications. It is acceptable to prescribe oral iron supplements. However, gastrointestinal side effects are very common and those lead to patient's intolerance as well as low patient's compliance. In those cases, as well as in severe anemia it is recommended to give iron sucrose. This drug is administered intravenously is effective to treat iron deficiency anemia with a minimal adverse effect profile. The two methods of giving iron sucrose is (1) to give I.V 200 mg iron sucrose 2-3 times/week or (2) to give I.V 500 mg iron sucrose once a week In the present study we aim to compare between the efficacy of those 2 protocols.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Iron deficiency anemia
* Intolerance or low compliance for oral iron

Exclusion Criteria:

* Known allergy for iron supplements
* Anemia not due to iron deficiency
* Acute infection
* Liver failure or viral hepatitis
* Thalassemia or hemoglobinopathies
* Asthma
* Multiple pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
The change between the hemoglobin level at randomization and the hemoglobin level at the time of delivery | from randomization to delivery
  Hemoglobin levels will be obtained at the beginning of the study and around delivery
Women's satisfaction from the protocol treatment according to the VAS (visual analog scale) | The day after delivery

SECONDARY OUTCOMES:
Type and rate of adverse events | Up to 30 weeks
The rate of patients who discontinued treatment | Up to 30 weeks
The weekly change in hemoglobin level, ferritin, serum iron, transferrin, MCV, iron saturation and reticolocyte count from randomization | Up to 4 weeks
The change in hemoglobin level, ferritin, serum iron, transferrin, MCV, iron saturation and reticolocyte count from the last dose of iron sucrose to delivery in 3 weeks intervals | Up to 30 weeks
The need for blood transfusion post partum | up to 4 days post partum
The need for iron sucrose administration post partum | up to 4 days post partum
The rate of anemia associated symptoms | From randomization and up to 30 weeks
The levels of neonatal hemoglobin, ferritin and bilirubin | up to 4 days post partum
The rate of neonatal polycythemia and need for phototherapy | up to 4 days post partum